CLINICAL TRIAL: NCT04939259
Title: A Comparative Clinical Investigation of Musician's Preference Between a General Listening Program and a New Music Rationale for Hearing Aids
Brief Title: A Comparative Clinical Investigation of Musician's Preference With Hearing Aids
Acronym: BF007-2101
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bernafon AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BF007-2101
Record Dates: First submitted 2021-06-08; First posted 2021-06-25 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: All participants will wear the new devices at the same time. They will have the general listening program and the new music program available in the same device. They will switch between the programs to make the comparison in multiple environments.
Who Masked: Participant
Masking Description: The order of the programs is blinded so that subjects don't know which slot (2 or 3) contains the music program or the general program. Slot 1 always has a general program for everyday speech understanding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Music Program (Experimental): The new hearing aid contains the new music program will be worn by all participants at the same time. The participants must switch between the two programs during use to make the comparison.
  Interventions: Device: New Music Program; Device: Standard Listening Program
- Standard Listening Program (Active Comparator): The new hearing aid also contains the standard listening program worn by all participants at the same time. The participants must switch between the two programs during use to make the comparison.
  Interventions: Device: New Music Program; Device: Standard Listening Program

INTERVENTIONS:
Device: New Music Program — A mini behind-the-ear hearing aid that amplifies sounds and directs them into the ear. The music program within the hearing aid will provide amplification specifically tuned for listening to music.
Device: Standard Listening Program — A mini receiver-in-the-ear hearing aid that amplifies sounds and directs them into the ear. The standard listening program within the hearing aid will provide amplification specifically tuned for listening to speech and daily general sounds in the environment.

SUMMARY:
For this study, Bernafon AG will carry out testing with participants with hearing loss to compare a dedicated music program to a general listening program. The Bernafon hearing aids used for the current study are CEmarked and will be released to the market in early 2022. The goal is to determine whether musicians will perceive a difference and prefer the music program over the default listening program in real-life situations. The devices will also be validated for performance before their release to the market.

DETAILED DESCRIPTION:
The intended use of hearing aids is to amplify sounds to compensate for hearing loss. The initial goal is to amplify speech and facilitate speech understanding especially in noise. Research shows that wireless hearing aids are efficacious for older adults , and in general, an increase in satisfaction and substantial benefits are characteristic for the wireless hearing aids brought to market during in the last decade.

Music is proven to enhance the lives of older people, but many people report a reduction in their ability to enjoy music with a hearing loss. Amplification can be used to overcome a hearing impairment and return the joy of music to those with hearing loss. However, for listening to music or particularly, for musicians that play an instrument, the hearing aid settings used for amplifying speech often have adverse effects on music.

Amplification and signal processing within hearing aids are designed to mainly improve speech understanding. It is possible to model the acoustical characteristics of speech because they are defined by the human vocal tract characteristics and the articulation speed. This acoustical model of speech is then used as a guideline for optimizing signal processing within the hearing aid. This approach has shown limitations in terms of perceived sound quality when listening to recorded or live music due to the characteristics of music which show more variations than speech in terms of frequency range, sound level, modulation, and dynamic range. These differences suggest that a specific listening program should be used when music is present in the listening environment. The need to offer a music program for musicians and music enthusiasts is also motivated by 1) the prevalence of hearing loss and associated audiological symptoms among musicians or music listeners exposed to high sound levels (and 2) the benefit (social, cognitive, and physical) of playing or listening to music especially for hearing impaired and seniors.

An optimization procedure based on the participation of the musician during the fitting procedure showed promising results in terms of preference when playing music and in discrimination thresholds of level, duration, and pitch. However, this procedure targets only musicians who actively play music and requires time, some specific knowledge, and the possibility to make the adjustments in the fitting room. A new fitting rationale dedicated to music was therefore developed and made available in the fitting software.

This new music rationale can be offered to any hearing aid user who wants an optimal listening experience when playing or listening to music (live, over a playback setup, or streaming from wireless device). The new music rationale is programmed based on the hearing loss and uses different gain shaping and kneepoints in the dynamic compression compared to the general listening program. Specific settings of signal processing features like directionality, noise reduction, or feedback cancellation are either turned off or set at a lower level than in the general listening program.

For this study, Bernafon AG will carry out testing with participants that are musicians with hearing loss to test the new music rationale. The current study will compare the standard listening program to the music program based on the new rationale. The Bernafon hearing aids used for the current study are CE- marked and the family of hearing aids have been on the market for almost one year. The hardware used for this test will be released in early 2022. The goal is to determine whether musicians will perceive a difference and prefer a music program over the general listening program when listening or playing music in real-life situations and to validate the performance of the hardware style before release to the market. The devices used for the trial are the Bernafon Alpha 9 mBTE and as the control device, the Bernafon Viron 9 miniRITE (MNR) behind-the-ear (BTE) hearing aids. The results of the trial will be used to examine differences in the benefit provided by the two programs as well as identify further optimization possibilities or new risks associated with the devices. Objective measures will be made with Real Ear Measures (REM) to verify the output of the hearing aids, and subjective differences will be measured with questionnaires, an adaptive music perception test, and a forced choice AB listening preference test.

All participants are hearing impaired persons that play an instrument. The trial will consist of a total of 2 appointments. For the field testing and the lab testing, the order of the test programs (music or standard) will be randomized. It is expected that the music program will perform better than the general listening program for perception and preference testing.

In summary, the primary goal of this study is to evaluate the performance of a music program based on a new rationale and to validate the performance of the devices before the release of a new style to the market.

ELIGIBILITY:
Inclusion Criteria:

* All classifications of hearing loss (sensorineural, conductive, mixed)

  * If the hearing loss is conductive or mixed it must be approved for amplification by a physician
  * All shapes of hearing loss (flat, sloping, reverse slope, notch)
  * Severity ranging from mild to severe
  * German speaking
  * Play a musical instrument
  * Both genders
  * Ages 18 and older
  * Ability and willingness to sign the consent form

Exclusion Criteria:

* Normal hearing

  * Contraindications for amplification
  * Active ear disease
  * Don't play an instrument
  * Inability to follow the procedures of the study due to language problems, psychological disorders, dementia, or other cognitive problems of the participant
  * A reduced mobility making them unable to attend weekly study appointments
  * A reduced ability to describe auditory impressions and the usage of the hearing aids
  * Uncooperative so that it is not possible to record a valid pure tone audiogram
  * A strongly reduced dexterity
  * Central hearing disorders
  * Bernafon employees
  * Family members of Bernafon employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
The number of patients that prefer the music program for listening to music over the standard listening program as reported in the questionnaire that asks patients to choose a program and state the reason why it was preferred. | 10 days
  A questionnaire will ask patients to choose between the music program and the standard listening program as their preferred program for listening to music. It is not a forced choice as they also have the option to choose "no preference." They are then asked to choose from a checkbox with a list of possible reasons for the preference as well as the ability to write in additional reasons.

SECONDARY OUTCOMES:
The number of patients that prefer the sound quality of the music program over the standard listening program measured with a forced choice A/B question on a touch screen. | 10 days
  Patients will listen to various styles of recorded music in the test booth while switching between hearing aid programs labelled as A and B to make a direct comparison. The test is a forced choice between A and B selected on a touch screen. Patients will not know which program is A and which is B. This will be based on the original randomization assigned to them at visit one.
The average level of decibels at which patients are able to discriminate the changes in pitch of recorded music samples as measured with a standardized test called the Adaptive Music Perception (AMP) test. | 0 days
  Patients will be tested in the sound booth with recorded music and make a forced choice between two pitch levels using the music program and using the standard listening program. The measurement scale is in decibels and a lower score signifies a better score. Patients must correctly identify four consecutive pitches before an average level is calculated.
The average level at which patients correctly repeat sentences presented in background noise using the standardized Gottingen Sentence Test (GOSA). | 10 days
  Recorded speech is presented in background noise using the standardized Gottingen Sentence Test (GOSA). The score is in signal-to-noise ratio with a lower score signifying a better answer. The sentences are presented at an adaptive level of the speech signal. The test is automated and changes the signal of the speech to maintain a 50% level of understanding.

OTHER OUTCOMES:
The number of patients with treatment-related adverse events as assessed by CTCAE v4.0. | 0 Days and 10 Days
  All adverse events will be collected at each appointment and assessed using the common terminology for AEs as described in the protocol. The treatment-related adverse events will be used as the measure to determine the safety of the device and whether there are new unexpected events related to the use of the device. The expected range of occurrences could vary from 0 to infinity, but only one new treatment-related adverse event would require a new risk assessment of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Simon, AuD, Principal Investigator — Bernafon AG
Locations (1):
- Bernafon AG, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
The anonymized data that is shared in the report will be made available to other researchers.